CLINICAL TRIAL: NCT00262873
Title: A Phase II Pilot Study of VELCADE in Patients With MDS
Brief Title: Bortezomib in Treating Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jane Liesveld, attending physician, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000449689; URCC-U20403; MILLENNIUM-i34103-042
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Myelodysplastic Syndromes
Keywords: previously treated myelodysplastic syndromes; refractory anemia with excess blasts; refractory anemia with ringed sideroblasts; refractory anemia; secondary myelodysplastic syndromes; de novo myelodysplastic syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib (Experimental)
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well bortezomib works in treating patients with myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of bortezomib, in terms of reduced cytopenia, in patients with myelodysplastic syndromes.
* Determine the safety and toxic effects of this drug in these patients.

Secondary

* Determine changes in marrow blast percentage or karyotypic profile in patients treated with this drug.

OUTLINE: This is an open-label study.

Patients receive bortezomib IV on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 1 year.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of myelodysplastic syndromes (MDS)
* Requires treatment or transfusion support for MDS, as indicated by 1 of the following:

  * Demonstrates transfusion or epoetin alfa dependence

    * Transfusion dependence is defined as requiring ≥ 2 units of packed RBCs within an 8-week period prior to study entry
  * Hemoglobin < 11g/dL on 2 separate occasions 2 weeks apart

    * No iron, cyanocobalamin (vitamin B_12), or folic acid deficiency or other causes of anemia
* Must have 1 of the following FAB subtypes:

  * Refractory anemia
  * Refractory anemia with ringed sideroblasts
  * Refractory anemia with excess blasts
  * Secondary MDS (if ≥ 3 years since active primary cancer)
* No chronic myelomonocytic leukemia
* Not refractory to platelet transfusion support (i.e., inability to maintain platelet count > 20,000/mm^3 with transfusion)
* No current acute myelogenous leukemia (e.g., > 30% blasts)

PATIENT CHARACTERISTICS:

Performance status

* Karnofsky 50-100%

Life expectancy

* At least 6 months

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin ≤ 2 mg/dL
* AST and ALT < 2 times upper limit of normal

Renal

* Creatinine clearance ≥ 30 mL/min

Cardiovascular

* No significant cardiovascular condition that would preclude study participation
* No uncontrolled hypertension

Pulmonary

* No significant pulmonary condition that would preclude study participation

Immunologic

* No serious concurrent infection

  * Active infections must be adequately treated with antibiotics prior to study entry
* No hypersensitivity to bortezomib, boron, or mannitol

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 4 weeks after completion of study treatment
* No peripheral neuropathy ≥ grade 2
* No uncontrolled seizure activity, as defined by no activity within the past year on stable anticonvulsant medications
* No other malignancy within the past 3 years except adequately treated basal cell skin cancer or carcinoma in situ of the cervix
* No endocrine, neurologic, or other systemic disease that would preclude study entry

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior allogeneic bone marrow transplantation
* Concurrent transfusion support allowed
* Concurrent epoetin alfa or darbepoetin alfa allowed if initiated before start of study therapy, dose is stable for ≥ 4 weeks, and dose is stable during study participation
* No concurrent platelet growth factor support
* No concurrent thalidomide

Chemotherapy

* No concurrent chemotherapy
* No concurrent hydroxyurea

Endocrine therapy

* Concurrent corticosteroids for chronic autoimmune or inflammatory condition allowed if initiated before start of study therapy and maintained on a stable or decreasing dose

Other

* Recovered from all prior therapies
* At least 4 weeks since prior MDS therapy, except epoetin alfa, darbepoetin alfa, filgrastim (G-CSF), pegfilgrastim (G-CSF), or transfusion support
* At least 30 days since prior investigational agents
* No prior bortezomib
* No other concurrent investigational agents
* No other concurrent therapy for MDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane L. Liesveld, MD, Study Chair — James P. Wilmot Cancer Center
Locations (1):
- James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Result] Liesveld JL, Rosell KE, Bechelli J, Lu C, Messina P, Mulford D, Ifthikharuddin JJ, Jordan CT, Phillips Ii GL. Proteasome inhibition in myelodysplastic syndromes and acute myelogenous leukemia cell lines. Cancer Invest. 2011 Aug;29(7):439-50. doi: 10.3109/07357907.2011.590567. PMID 21740082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 patients were screened for the study.
Pre-assignment Details: 15 patients did not meet study eligibility criteria.
Groups:
- Bortezomib: Bortezomib was given at a dose of 1.3 mg per meter squared on day 1, 4, 8, and 11 on a 21 day cycle. Up to 12 cycles were allowed. Response assessments were made after the 3rd, 6th and 12 cycles of therapy.
Period: Overall Study
Arm/Group | Bortezomib
Started | 8
Completed | 0
Not Completed | 8
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 69 [51 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Time Frame: For 21 days/course for up to 12 courses
Population: patients enrolled to receive study drug
Measure: Number; unit: participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 8
participants | 6

2. Primary Outcome: Number of Participants Who Experienced Cytopenias
Time Frame: 21 Days/course for up to 12 courses
Population: This data was not collected.
Arm/Group | Bortezomib
Number analyzed (Participants) | 0

3. Secondary Outcome: Interleukin 6 Levels in Serum
Description: interleukin-6 levels were measured by enzyme-linked immunosorbant assay ELISA in serum from participants exposed to bortezomib.
  Levels were measured at Day 0 and Day 14 of cycle 1 of the clinical trial.
Time Frame: day 14
Population: data was only available on 5 participants
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Bortezomib
Number analyzed (Participants) | 5
pg/ml
  pre bortezomib | 6.8 (1.7)
  post bortezomib | 8.6 (3.3)
Statistical Analysis 1: Comparison: Bortezomib; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

4. Secondary Outcome: Vascular Endothelial Growth Factor (VEGF) Levels in Serum
Description: VEGF levels were measured by ELISA (R&DSystems) in serum from participants exposed to bortezomib. Levels were measured at Day 0 and Day 14 of cycle 1 of the clinical trial.
Time Frame: day 14
Population: data was only available on 5 participants
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Bortezomib
Number analyzed (Participants) | 5
pg/ml
  pre bortezomib | 402 (105)
  post bortezomib | 254 (69)
Statistical Analysis 1: Comparison: Bortezomib; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

5. Secondary Outcome: Average Percentage of Light Density Cells in Apoptosis
Description: The CD34+ fraction of light density marrow obtained from patients at baseline and while receiving bortezomib were assessed through measurement of Annexin V (assay obtained form R&D Systems) and by flow cytometry analysis.
Time Frame: day 14
Population: marrow samples were not available on all participants at baseline
Measure: Mean (Standard Deviation); unit: percentage of apoptotic cells
Arm/Group | Bortezomib
Number analyzed (Participants) | 5
percentage of apoptotic cells
  pre bortezomib | 6.68 (2.67)
  post bortezomib | 11.37 (3.73)
Statistical Analysis 1: Comparison: Bortezomib; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

6. Secondary Outcome: Average Number of Colony Forming Unit-granulocyte-macrophages in Bone Marrow
Description: Colony forming unit-granulocyte-macrophage (CFU-GM) progenitors, erythroid burst forming units (BFU-E), and leukemia colony forming units (CFU-L) were measured at day 0 and day 14 of cycle 1. Five × 10(4) light density cell for granulocyte-macrophage colony forming unit (CFU-GM) or erythroid burst forming unit (BFU-E) assays were plated in 0.9% methylcellulose, 30% FCS, 2 mmol/L L-glutamine, 10-4 mol/L β-mercaptoethanol, and 1% BSA with 3U/ml human erythropoietin, 10 ng/ml GM-CSF, 10 ng/ml IL-3, and 50 ng/ml stem cell factor (SCF) (c-kit ligand). For leukemia colony forming units (CFU-Ls), the plating mixture was comparable with the exception that the cytokines utilized were 4 U/ml erythropoietin, 10 ng/ml GM-CSF, 10 ng/ml IL-3, 100 ng/ml c-kit ligand, and 100 ng/ml Flt3 ligand. The methylcellulose mixture and associated reagents were purchased from Stem Cell Technologies (Vancouver, BC). Colonies were scored at Day 14 and were defined as > 20 grouped cells.
Time Frame: day 14
Population: baseline marrow samples were available only 5 participants
Measure: Mean (Standard Deviation); unit: number of colonies per 50000 cell plated
Arm/Group | Bortezomib
Number analyzed (Participants) | 5
number of colonies per 50000 cell plated
  pre bortezomib | 16.1 (12.8)
  post bortezomib | 28.6 (25.8)

7. Secondary Outcome: Average Number of Erthroid Burst Forming Units in Bone Marrow
Description: as for outcome 6
Time Frame: day 14
Population: analysis was performed on only four participants
Measure: Mean (Standard Deviation); unit: number of colonies per 50000 cell plated
Arm/Group | Bortezomib
Number analyzed (Participants) | 4
number of colonies per 50000 cell plated
  pre bortezomib | 14.75 (14.98)
  post bortezomib | 14.75 (25.51)

8. Secondary Outcome: Average Number of Leukemia Forming Units in Bone Marrow
Description: as for outcome 6
Time Frame: day 14
Population: baseline bone marrow was only available on 5 participants
Measure: Mean (Standard Deviation); unit: number of colonies per 50000 cell plated
Arm/Group | Bortezomib
Number analyzed (Participants) | 5
number of colonies per 50000 cell plated
  pre bortezomib | 27.65 (25.15)
  post bortezomib | 54.28 (59.16)

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Bortezomib
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib (N=8)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib (N=8)
Hypotension (Cardiac disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4)
Fever (Infections and infestations) | 1 (1)
Low Platelets (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
All study visits were completed and the trial concluded normally for the limited number of enrolled participants; therefore, the study was considered to have been completed. However, the study is under-powered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No